CLINICAL TRIAL: NCT01631175
Title: Establishment of an Indication-based Identification and Psychosocial Treatment of Orthopedic Cancer Patients Suffering From Psychosocial Stress
Brief Title: Indication-based Identification and Psychosocial Treatment of Orthopedic Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Lenze-2011
Record Dates: First submitted 2012-06-20; First posted 2012-06-29 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Psychological Distress
Keywords: sarcoma; distress; tumor; quality of life; cancer
MeSH Terms: conditions — Sarcoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (PO-Bado, FBK-R10, PHQ) Active Comparator (Experimental)
  Interventions: Behavioral: psychosocial treatment

INTERVENTIONS:
Behavioral: psychosocial treatment — psychosocial treatment, verbal therapy, relaxation exercises
  Other Names: PO-Bado; Patient Health Questionaire; Questionaire for Psychosocial Burden of Cancer Patients

SUMMARY:
Aim of this study is to develop and establish an indication-based algorithm for identifying particular stress patterns of patients with initial diagnosis of a sarcoma or a metastatic bone disease. A further aim was the establishment of an adequate psychosocial treatment within the clinical workday routine to support coping with illness and treatment.

DETAILED DESCRIPTION:
Aim of this study is to develop and establish an indication-based algorithm for identifying particular stress patterns of patients with initial diagnosis of a sarcoma or a metastatic bone disease. A further aim was the establishment of an adequate psychosocial treatment within the clinical workday routine to support coping with illness and treatment.

Methods:

Patients with histologically assured sarcoma or metastatic bone disease are psycho-oncologically screened by a common cancer specific expert rating scale (PO-Bado: Basic Documentation for Psycho-Oncology, 6 items) at the time of admission before tumor resection. In the same line patients were asked to answer two standardized self-rating questionaires, namely the FBK-R10 (Questionaire for Psychosocial Burden of Cancer Patients, 10 items) and a modified form of the PHQ (Patient Health Questionaire, 2 items) to assess patients' burden of disease as well as the presence of depressive mood. Cancer patients exceeding a defined critical PO-Bado cut-off value (a minimum of 2 items scoring 3 or 1 item scoring 4) are expected to require psychosocial support and a psychosocial consultation/co-treatment iss initiated.

To evaluate short-term effects of the psycho-social treatment the cancer-specific screening is repeated (PO-Bado, FBK-R10, PHQ) before discharge from the hospital. All diagnostic findings as well as a specific recommendation for the continuing treatment are integrated into the orthopedic discharge letter. Furthermore, all findings are shown and factored for decision making within the interdisciplinary musculoskeletal tumor board. For appraisal of treatment-based long-term effects the psycho-oncological screening is repeated within the orthopedic aftercare examinations 3 and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18
* initial diagnosis of a histologically assured sarcoma or metastatic bone disease

Exclusion Criteria:

* age younger than 18
* benign tumors
* patients with known sarcoma or metastatic bone disease
* patients with known other tumors
* fundamental neurological and psychiatric disorders
* prisoners
* patients with guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Psychooncological Basic Documentation (PO-BADO) | 0,6,12 month
  The PO-BADO is a cancer-specific screening instrument. It enables clinical staff to screen cancer patients for the need of psycho-oncological support as well as to document and assess psychosocial stress. The PO-Bado has been psychometrically evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Lenze, MD, Principal Investigator — Department for Orthopedics and Orthopedic Sports Medicine, Klinikum rechts der Isar der TU München
Locations (1):
- Department of Orthopedics and Orthopedic Sports Medicine, Munich, Bavaria, Germany

REFERENCES:
- [Background] Herschbach P, Book K, Brandl T, Keller M, Marten-Mittag B. The Basic Documentation for Psycho-Oncology (PO-Bado): an expert rating scale for the psychosocial experience of cancer patients. Onkologie. 2008 Nov;31(11):591-6. doi: 10.1159/000162287. Epub 2008 Oct 27. PMID 19145091